CLINICAL TRIAL: NCT00081354
Title: Barrett's Esophagus Early Detection Study
Brief Title: Early Detection of Barrett's Esophagus
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040155; 04-C-0155; NCT00899106 (obsolete NCT alias)
Record Dates: First submitted 2004-04-09; First posted 2004-04-09 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Barrett's Esophagus
Keywords: Biopsy Tissue; Barrett Esophagus; Gastroesophageal Reflux Disease; GERD; Dysphagia; Swallowing Difficulty
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

GROUPS / COHORTS (2):
- Barrett's esophagus: Barrett's esophagus
- Controls negative for Barrett's esophagus: Controls negative for Barrett's esophagus

SUMMARY:
Background:

The incidence rate for esophageal adenocarcinoma (EAC) has risen 10% per year over the past two decades and is the most rapidly increasing cancer in the U.S.

Barrett's esophagus (BE), a metaplastic change from the normal squamous esophageal epithelium to a specialized intestinal-type columnar mucosa, increases the risk of EAC by 30-125, and is considered a precursor lesion for EAC.

Individuals diagnosed with BE are currently entered into endoscopic surveillance programs to look for dysplasia or EAC. However, only 5% of subjects diagnosed with EAC have a previous diagnosis of BE or have been part of a surveillance program, so alternative screening methods are needed.

Objectives:

The primary goal of this project is to identify a practical blood-based biomarker(s) that can be used as a screening test to determine who has BE and who does not.

Secondary goals of the project are to characterize germ-line and tissue biomarkers associated with BE, and to compare biomarkers in non-BE patients with and without GERD.

Tertiary goals are to explore associations between biomarkers in blood or tissue and progression from BE to dysplasia or EAC, and to assess the stability of proteomic patterns over time.

Eligibility:

This study will be conducted among patients in the Barrett's Esophagus Registry (currently with 206 registrants) established at the National Naval Medical Center (NNMC) in Bethesda beginning in 1992, as well as a comparison group of approximately 600 matched non-BE patients endoscoped in the GI clinic at NNMC for other conditions.

Design:

Blood and tissue samples will be collected as well as questionnaire data on risk factors and medications as well as GERD.

Data analyses will be based primarily on laboratory testing of newly collected esophageal biopsies, brush samples, and blood samples, but secondarily will also include use of archival tissue biopsy samples.

Follow up of BE Registry patients will include standard periodic surveillance endoscopies, additional blood samples, and ascertainment of disease status (i.e., progression).

To distinguish BE versus non BE-patients in this case-control study, we will:

assess predictability of BE status from serum proteomic patterns;

characterize esophageal biopsies and brush samples for selected DNA alterations, RNA expression, and proteomic profiles;

genotype patients for selected polymorphisms potentially associated with BE;

compare blood and tissue biomarkers in non-BE patients with and without GERD;

explore the association of biomarkers with progression from BE to dysplasia or EAC;

assess proteomic pattern stability over time in BE patients.

DETAILED DESCRIPTION:
Background:

The incidence rate for esophageal adenocarcinoma (EAC) has risen 10% per year over the past two decades and is the most rapidly increasing cancer in the U.S.

Barrett's esophagus (BE), a metaplastic change from the normal squamous esophageal epithelium to a specialized intestinal-type columnar mucosa, increases the risk of EAC by 30-125 fold (1), and is considered a precursor lesion for EAC.

Individuals diagnosed with BE are currently entered into endoscopic surveillance programs to look for dysplasia or EAC. However, only 5% of subjects diagnosed with EAC have a previous diagnosis of BE or have been part of a surveillance program, so alternative screening methods are needed.

Objectives:

The primary goal of this project is to identify a practical blood-based biomarker(s) that can be used as a screening test to determine who has BE and who does not.

Secondary goals of the project are to characterize germ line and tissue biomarkers associated with BE, and to compare biomarkers in non-BE patients with and without GERD.

Tertiary goals are to explore associations between biomarkers in blood or tissue and progression from BE to dysplasia or EAC, and to assess the stability of proteomic patterns over time.

Eligibility:

This study will be conducted among patients in the Barretts Esophagus Registry (currently with 206 registrants) established at the National Naval Medical Center (NNMC) in Bethesda beginning in 1992 as well as comparison group of approximately 600 matched non-BE patients endoscoped in the GI clinic at NNMC for other conditions.

Design:

Blood and tissue samples will be collected as well as questionnaire data on risk factors and medications as well as GERD.

Data analysis will be based primarily on laboratory testing of newly collected esophageal biopsies, brush samples, and blood samples, but secondarily will also include use of archival tissue biopsy samples.

Follow-up of BE Registry patients will include standard periodic surveillance endoscopies, additional blood samples, and ascertainment of disease status (i.e, progression).

To distinguish BE versus non-BE patients, we will: (1) assess predictability of BE status from serum proteomic patters; (2) characterize esophageal biopsies and brush samples for selected DNA alterations, RNA expression, and proteomic profiles; (3) genotype patients for selected polymorphisms potentially associated with BE; (4) compare blood and tissue biomarkers in non-BE patients with and without GERD; (5) explore the association of biomarkers with progression from BE to dysplasia or EAC; and (6) assess proteomic pattern stability over time in BE patients.

ELIGIBILITY:
* INCLUSION CRITERIA

Inclusion criteria for EGD in this study include:

Greater than or equal to 18 years of age, and

presence of GERD or GERD-like symptoms, or

presence of BE, or

dysphagia, or

anemia, or

gastrointestinal bleeding, or

presence of other conditions (e.g., dyspepsia) that merit endoscopic evaluation.

EXCLUSION CRITERIA

Exclusion criteria for EGD in this study include:

severe pulmonary or cardiac disease, or

pregnancy, or

refusal, or

inability or refusal to give consent, or

age less than 18 years or participation in NNMC Barrett's esophagus cryotherapy protocol, or

malignancy other than nonmelanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: National Naval Medical Center (NNMC) in Bethesda
Sampling Method: Non-Probability Sample
Enrollment: 737 (Actual)
Dates: Start 2004-04-06 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Case Control | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Cook, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Naval Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gerson LB, Shetler K, Triadafilopoulos G. Prevalence of Barrett's esophagus in asymptomatic individuals. Gastroenterology. 2002 Aug;123(2):461-7. doi: 10.1053/gast.2002.34748. PMID 12145799
- [Background] di Pietro M, Lao-Sirieix P, Boyle S, Cassidy A, Castillo D, Saadi A, Eskeland R, Fitzgerald RC. Evidence for a functional role of epigenetically regulated midcluster HOXB genes in the development of Barrett esophagus. Proc Natl Acad Sci U S A. 2012 Jun 5;109(23):9077-82. doi: 10.1073/pnas.1116933109. Epub 2012 May 17. PMID 22603795
- [Background] Yasui Y, Pepe M, Thompson ML, Adam BL, Wright GL Jr, Qu Y, Potter JD, Winget M, Thornquist M, Feng Z. A data-analytic strategy for protein biomarker discovery: profiling of high-dimensional proteomic data for cancer detection. Biostatistics. 2003 Jul;4(3):449-63. doi: 10.1093/biostatistics/4.3.449. PMID 12925511
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-C-0155.html